CLINICAL TRIAL: NCT05409872
Title: Effects of Vitamin D, Epigallocatechin Gallate, Vitamin B6, and D-Chiro-inositol Combination on Uterine Fibroids: a Randomized Controlled Trial
Brief Title: Effects of Vitamin D, Epigallocatechin Gallate, Vitamin B6, and D-Chiro-inositol Combination on Uterine Fibroids
Acronym: DEFIB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Prof., Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEFIB
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Leiomyoma, Uterine
Keywords: Leiomyoma, Uterine; Epigallocatechin gallate; Vitamin D; D-Chiro-inositol; Vitamin B6
MeSH Terms: conditions — Leiomyoma | interventions — Vitamin D; Vitamin B 6

STUDY DESIGN:
Intervention Model Description: Randomized (1:1) double-blind, single-center controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination of Epigallocatechin gallate, vitamin D, vitamin B6, and D-Chiro-inositol (Experimental): The subject takes a combination of 333.35 mg of green tea extract (150 mg of Epigallocatechin gallate), 25 mg of D-Chiro-inositol, 25 mcg of Vitamin D, and 5 mg of Vitamin B6 twice a day for three months.
  Interventions: Dietary Supplement: Combination of Epigallocatechin gallate, vitamin D, vitamin B6, and D-Chiro-inositol
- Placebo (Placebo Comparator): The subject takes the placebo twice a day for three months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Combination of Epigallocatechin gallate, vitamin D, vitamin B6, and D-Chiro-inositol — The subject takes a combination of 333.35 mg of green tea extract (150 mg of Epigallocatechin gallate), 25 mg of D-Chiro-inositol, 25 mcg of Vitamin D, and 5 mg of Vitamin B6 twice a day for three months.
  Arms: Combination of Epigallocatechin gallate, vitamin D, vitamin B6, and D-Chiro-inositol
Other: Placebo — The subject takes the placebo twice a day for three months.
  Arms: Placebo

SUMMARY:
Randomized (1:1) double-blind, single-center controlled trial to evaluate the efficacy of 3 months of treatment with Epigallocatechin gallate, vitamin D, D-Chiro-inositol, and vitamin B6 on symptoms related to uterine fibroids

DETAILED DESCRIPTION:
A randomized controlled trial aimed to evaluate the efficacy of a combination of Epigallocatechin gallate, vitamin D3, D-Chiro-inositol, and vitamin B6 as a treatment for uterine fibroids. The clinical study is double-blind, neither patients nor investigators know whether the subject receives the combination of Epigallocatechin gallate, vitamin D, D-Chiro-inositol, and vitamin B6 or the placebo. After 3 months of treatment, changes in symptoms associated with uterine fibroids, quality of life, and ultrasounds characteristics are compared between the two treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Women with multiple fibroids or single fibroma with a diameter ≥ 4 cm who are candidates for hysterectomy.
* Women with multiple fibroids or single fibroma with a diameter ≥ 4 cm who are candidates for myomectomy / uterine arterial embolization.
* Women with multiple fibroids or single fibroma with a diameter ≥ 4 cm who are candidates for treatment with magnetic resonance (MR)-guided Focused Ultra-Sound (MrgFUS).

Exclusion Criteria:

* Pregnancy.
* Breastfeeding.
* Smoking.
* Suspected malignancy.
* Patients who have undergone medical treatment for uterine fibroids within the previous three months.
* Patients allergic to the components of the product or placebo under study.
* Patients who refuse to provide informed consent to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms related to uterine fibromatosis (UFS-QoL questionnaire) | After 3 months of treatment
  Symptoms related to uterine fibromatosis assessed with the eight symptom questions of the Fibroid Symptom and Quality of Life (UFS-QoL) questionnaire. Score: min 8 - max 40, with higher scores meaning worse outcome.

SECONDARY OUTCOMES:
The proportion of patients who refuse surgery due to regression of symptoms. | After 3 months of treatment
  The proportion of patients who refuse surgery due to regression of symptoms.
Volume of the larger fibroid | After 3 months of treatment
  Volume of the larger fibroid assessed by transvaginal ultrasound
Quality of life (UFS-QoL questionnaire) | After 3 months of treatment
  Quality of life assessed with the 29 health-related quality of life questions of the Fibroid Symptom and Quality of Life (UFS-QoL) questionnaire. Score: min 29 - max 145, with higher scores meaning worse outcome.
The total score obtained in the Menstrual assessment chart | After 3 months of treatment
  The total score obtained in the Menstrual assessment chart. Score: min 0 - N/A max, with higher scores meaning worse outcome.
The total score obtained in the Pad test | After 3 months of treatment
  The total score obtained in the Pad test. Score: min 0 - N/A max, with higher scores meaning worse outcome.
Proportion of patients who reported side effects or who stopped taking the treatment | After 3 months of treatment
  Proportion of patients who reported side effects or who stopped taking the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, MD, PhD, Principal Investigator — AOUI Verona - University of Verona; Simone Garzon, MD, Principal Investigator — AOUI Verona - University of Verona; Pier Carlo Zorzato, MD, Principal Investigator — AOUI Verona - University of Verona
Locations (1):
- AOUI Verona - University of Verona - Department of Obstetrics and Gynecology, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baird DD, Hill MC, Schectman JM, Hollis BW. Vitamin d and the risk of uterine fibroids. Epidemiology. 2013 May;24(3):447-53. doi: 10.1097/EDE.0b013e31828acca0. PMID 23493030
- [Background] Roshdy E, Rajaratnam V, Maitra S, Sabry M, Allah AS, Al-Hendy A. Treatment of symptomatic uterine fibroids with green tea extract: a pilot randomized controlled clinical study. Int J Womens Health. 2013 Aug 7;5:477-86. doi: 10.2147/IJWH.S41021. eCollection 2013. PMID 23950663
- [Background] Porcaro G, Santamaria A, Giordano D, Angelozzi P. Vitamin D plus epigallocatechin gallate: a novel promising approach for uterine myomas. Eur Rev Med Pharmacol Sci. 2020 Mar;24(6):3344-3351. doi: 10.26355/eurrev_202003_20702. PMID 32271452
- [Background] Zhang D, Al-Hendy M, Richard-Davis G, Montgomery-Rice V, Rajaratnam V, Al-Hendy A. Antiproliferative and proapoptotic effects of epigallocatechin gallate on human leiomyoma cells. Fertil Steril. 2010 Oct;94(5):1887-93. doi: 10.1016/j.fertnstert.2009.08.065. Epub 2009 Oct 12. PMID 19819432